CLINICAL TRIAL: NCT03285776
Title: Reliability and Validity of a Computerized Tool to Assess Proprioception Among Children With Coordination Disorders
Status: Completed | Type: Observational
Sponsor: Jay Zuckerman (Other)
Responsible Party: Sponsor-Investigator, Jay Zuckerman, Developmental doctor and director of the Children's Development Center, Meir Medical Center
Organization: Meir Medical Center (Other)
Other Study IDs: MMC170038-17kCTIL
Record Dates: First submitted 2017-09-10; First posted 2017-09-18 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Developmental Coordination Disorder; Developmental Dyspraxia; Clumsy Child Syndrome
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Children with coordination disorder between the ages of 5 to 7 years.
- control group: children with typical development between the ages of 5 to 7 years.

SUMMARY:
Coordination disorders are common among children that arrive to child development services. Children with coordination disorders have impaired proprioceptive sensation and motor planning. It is important to carry out a comprehensive assessment of these children in order to design an appropriate and effective treatment. There is a lack of an objective and standard assessment tools for proprioception and motor planning. Technology based assessment tools might offer a solution, as they enable automated and accurate measurement. The purpose of this study is to examine the validity and reliability of a new diagnostic computerized kit, which was developed for assessment of proprioception and motor planning among children with coordination disorders. The hypothesis includes:

1. Examine the construct validity of the new diagnostic computerized kit (the known group procedure). Whether there is a difference in the outcomes between children with typical development and children with coordination disorders.
2. Examine the construct validity of the new diagnostic computerized kit outcomes - correlation with the following associated variables: (a) motor skills; (b) sensory function; (c) participation in daily activities.
3. Examine of test-retest reliability of the new diagnostic computerized kit. Whether the outcomes are stable in repeated measurements.

The participants will include fifty children between the ages of 5 to 7 years: 25 children with coordination disorders (study group), and 25 children with typical development (control group).

Each child will arrive for an evaluation meeting that includes: (a) the new diagnostic computerized kit; (b) standard and routine tests for motor skills (Movement Assessment Battery for Children-2-MABC-2, and two sub-test of the Beery-Buktenica developmental test of visual-motor integration- Beery VMI). In addition, the children's parents will complete two questionnaires: (a) Sensory Processing Measurement (SPM) for sensory function assessment; (b) Participation in Childhood Occupations Questionnaire (PICO-Q) for daily participation assessment. After two weeks, ten children from the control group will be evaluated once again by the new diagnostic computerized kit for examine test-retest reliability.

DETAILED DESCRIPTION:
Coordination disorders are common among children that arrive to child development services. Children with coordination disorders have impaired proprioceptive sensation and motor planning. It is important to carry out a comprehensive assessment of these children in order to design an appropriate and effective treatment. There is a lack of an objective and standard assessment tools for proprioception and motor planning. Technology based assessment tools might offer a solution, as they enable automated and accurate measurement. The purpose of this study is to examine the validity and reliability of a new diagnostic computerized kit, which was developed for assessment of proprioception and motor planning among children with coordination disorders.

The new diagnostic computerized kit consists a computerized thumb- fingers matching test (for proprioception).

The hypothesis includes:

1. Examine the construct validity of the new diagnostic computerized kit (the known group procedure). Whether there is a difference in the outcomes between children with typical development and children with coordination disorders.
2. Examine the construct validity of the new diagnostic computerized kit outcomes - correlation with the following associated variables: (a) motor skills; (b) sensory function; (c) participation in daily activities.
3. Examine of test-retest reliability of the new diagnostic computerized kit. Whether the outcomes are stable in repeated measurements.

The participants will include fifty children between the ages of 5 to 7 years: 25 children with coordination disorders (study group) in a waiting list for an occupational therapy evaluation (in Orlansky Children's Development Center, Dan -Petah Tikva Region, Clalit Health Services), and 25 children with typical development (control group).

The participants will be recruited by a convenience sample. Participation in the study will be offered by telephone to parents of children who may meet the inclusion /exclusion criteria. For the study group the recruitment will be to children in a waiting list for an occupational therapy evaluation (in Orlansky Children's Development Center). For the control group, the recruitment will be by a snowball sample (a friend brings a friend), through acquaintances of the investigators. Children whose parents agree to participate in the study will attend one meeting, accompanied by at least one parent. At the beginning of the meeting, the parents will receive a detailed explanation about the purpose and the study process. The new diagnostic computerized kit will be presented and explained how to use it. Parents will be assured total privacy. In addition, parents of children from the study group will be told that their child's medical record will be used to ensure inclusion and exclusion criteria. Parents who express their consent to participate in the study will sign an informed consent form and then complete a demographic questionnaire and a screening questionnaire. Children that will be find suitable for the study will Be evaluated by: (a) the new diagnostic computerized kit; (b) standard and routine tests for motor skills (Movement Assessment Battery for Children-2-MABC-2, and two sub-test of the Beery-Buktenica developmental test of visual-motor integration- Beery VMI). In addition, the children's parents will complete two questionnaires: (a) Sensory Processing Measurement (SPM) for sensory function assessment; (b) Participation in Childhood Occupations Questionnaire (PICO-Q) for daily participation assessment. After two weeks, ten children from the control group will be evaluated once again by the new diagnostic computerized kit for examine test-retest reliability.

Analysis of the data will be done using the SPSS version 32. Descriptive statistics will be used for description of the population and the variables. Shapiro-wilks test will be used to examine the type of distribution of the dependent variables. According to the type of distribution will use t-test for two independent samples or Mann-Whitney test to examine the differences between groups (hypothesis 1). Pearson Correlation Coefficient test or Spearman's Rank Correlation Coefficient test will be used to examine correlation between the outcomes of the assessment tools (hypothesis 2 and 3). The significance level for all the statistical tests will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-7, insured by "Clalit Health Services", and their parents. Inclusion into groups will be done according to the DCDQ'07 Developmental Questionnaire (DCDQ'07).
* Inclusion to study group: children in a waiting list for an occupational therapy evaluation due to difficulties in fine or gross motor difficulties in performing daily activities as self-treatment, Play and recreation, and suspicion of developmental delay and DCD. children are able to communicate and understand instructions in Hebrew, and their parents know the Hebrew language at the level of reading and writing. A score of 15-46 indicating DCD or suspected DCD in the DCDQ'07 questionnaire.
* Inclusion into control group: healthy children with a typical development who are able to communicate and understand Hebrew instructions, and whose parents know the Hebrew language at the level of reading and writing. A score of 47-75 indicates that there is no DCD in the DCDQ'07 questionnaire.

Exclusion Criteria:

* Children with developmental syndromes such as autism, cerebral palsy, orthopedic or neurological diseases, including sensory systems, such as impaired vision, will not be included in the study (according to parents' questioning, if no information will be available in the medical record). Children who study in special education frames (according to parental questioning) will not be included in the study. Children who have previously been treated in occupational therapy will not included.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants will include fifty children between the ages of 5 to 7 years:
  the study group - 25 children in a waiting list for an occupational therapy evaluation (in Orlansky Children's Development Center, Dan -Petah Tikva Region, Clalit Health Services), the control group - 25 children with typical development.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Total time- outcome of the new diagnostic computerized kit - computerized thumb fingers matching test. | Time duration for this test is 5 minutes.
  Time is one of the outcome measures of the computerized thumb fingers matching test, that is measured in a ratio scale.
Standard Deviation (SD) of touch time- outcome of the new diagnostic computerized kit - computerized thumb fingers matching test. | Time duration for this test is 5 minutes.
  Standard Deviation (SD) of touch time is one of the outcome measures of the computerized thumb fingers matching test, that is measured in a ratio scale by sensors of the touches.
Correct sequence- outcome of the new diagnostic computerized kit - computerized thumb fingers matching test. | Time duration for this test is 5 minutes.
  Correct sequence is one of the outcome measures of the computerized thumb fingers matching test, that is measured in a ratio scale by sensors of the touches.

SECONDARY OUTCOMES:
Visual-motor integration outcome of the Beery-Buktenica developmental test of visual-motor integration (Beery VMI). | Time duration for this test is 10 minutes. only one time point
  Visual-motor integration grade is measured in a ratio scale from the Beery VMI test.
Motor coordination outcome of the Beery-Buktenica developmental test of visual-motor integration (Beery VMI). | Time duration for this test is 5 minutes. only one time point
  Motor coordination grade is measured in a ratio scale from the Beery VMI test.
Physical awareness outcome of the Sensory Processing Measurement (SPM). | Time duration for this questionaire is 20 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Balance and movement outcome of the Sensory Processing Measurement (SPM) . | Time duration for this questionaire is 20 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Planning and ideation outcome of the Sensory Processing Measurement (SPM). | Time duration for this questionaire is 20 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Total sensory systems outcome of the Sensory Processing Measurement (SPM). | Time duration for this questionaire is 20 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Difficulty in performance outcome of the Participation in Childhood Occupations Questionaire (PICO-Q). | Time duration for this questionaire is 15 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Frequency of performance outcome of the Participation in Childhood Occupations Questionaire (PICO-Q). | Time duration for this questionaire is 15 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Enjoyment outcome of the Participation in Childhood Occupations Questionaire (PICO-Q). | Time duration for this questionaire is 15 minutes. only one time point
  Questionaire for the parents that is measured in a Likert scale.
Movement Assessment Battery for Children-2 (MABC-2)- general grade. | Time duration for this test is 30 minutes. only one time point
  General grade of the subject's motor performance, that is measured in a ratio scale from the MABC-2.
Balance outcome of the Movement Assessment Battery for Children-2 (MABC-2). | Time duration for this test is 10 minutes. only one time point
  Balance grade is measured in a ratio scale from the MABC-2.
Ball skills outcome of the Movement Assessment Battery for Children-2 (MABC-2). | Time duration for this test is 10 minutes. only one time point
  Ball skills grade is measured in a ratio scale from the MABC-2.
Fine manual skills outcome of the Movement Assessment Battery for Children-2 (MABC-2). | Time duration for this test is 10 minutes. only one time point
  Fine manual skills grade is measured in a ratio scale from the MABC-2.

CONTACTS AND LOCATIONS:
Overall Officials: jay zuckerman, DR, Principal Investigator — Israel: Clalit Health Services
Locations (1):
- Orlansky,Clalit Health Services, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided